CLINICAL TRIAL: NCT06113874
Title: The Influence of Desensitizing Agent on Postoperative Sensitivity in Posterior Composite Restoration: A Randomized Controlled Clinical Trial
Brief Title: The Influence of Desensitizing Agent on Postoperative Sensitivity in Posterior Composite Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 7/22
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — gluma desensitizer

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Composite with Hurriseal desensitizer (Experimental)
  Interventions: Other: Hurriseal desensitizer
- Composite with Gluma Desensitizer (Active Comparator)
  Interventions: Other: Gluma desensitizer
- Composite without desensitizer (No Intervention)

INTERVENTIONS:
Other: Hurriseal desensitizer — Patients will receive Hurriseal desensitizing agent and universal bond and composite.
  Cavities will be restored with light-cured composite resin following the application of bonding agent.
  Arms: Composite with Hurriseal desensitizer
Other: Gluma desensitizer — Patients will receive Gluma desensitizing agent and universal bond and composite.
  Cavities will be restored with light-cured composite resin following the application of bonding agent.
  Arms: Composite with Gluma Desensitizer

SUMMARY:
This study aims to investigate the influence of desensitizing agents on reducing post-operative sensitivity in posterior composite.

ELIGIBILITY:
Inclusion Criteria:

* Patients having active primary class I carious lesions on vital molar teeth either in the middle or the inner third of dentin in the three quadrants of each patients.
* Teeth having a positive reaction to vitality test (cold test), no signs of pulp inflammation, or spontaneous pain before treatment.
* Preoperative radiographic record of the carious lesions.
* Buccolingual width is no more than half the inter-cuspal distance

Exclusion Criteria:

* Excessive tooth wear due to clenching or abnormal habits.
* Patients with direct occlusal contact by antagonist cusp (traumatic occlusion).
* Patients with periodontal or gingival disease.
* Patients using analgesics and/or anti-inflammatory medicine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity assessment | up to 12 months
  Air spray will be applied from a 2-mm distance on to the occlusal for 3 seconds. The severity of patients' pain/sensitivity will be recorded using (0-10) numerical rating scale. The score will be ranged from 0 (No pain) to 10 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Nessrin Magdy, BDS, Principal Investigator — Alexandria University; Waleed El-Mahy, PhD, Study Director — Alexandria University; Rania R Afifi, PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt